CLINICAL TRIAL: NCT00001381
Title: A Phase I Trial Using Suramin to Treat Superficial Transitional Cell Carcinoma of the Bladder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940098; 94-C-0098
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Bladder Neoplasms; Carcinoma, Transitional Cell
Keywords: Adult; Intravesical Chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Suramin

INTERVENTIONS:
Drug: suramin

SUMMARY:
Patients with superficial transitional cell carcinoma of the bladder will be treated with intravesical suramin in a phase I dose escalating study. The toxicity of suramin administered in this fashion will be evaluated.

DETAILED DESCRIPTION:
Patients with superficial transitional cell carcinoma of the bladder will be treated with intravesical suramin in a phase I dose escalating study. The toxicity of suramin administered in this fashion will be evaluated.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically confirmed superficial transitional cell carcinoma of the bladder pathologically staged as Tis, Ta, or T1. Visible tumors at time of treatment not required. No metastatic disease or muscle invasion.

Clinically useful pretreatment bladder function required.

No significant prostatic obstructive symptoms associated with impaired or incomplete bladder emptying.

No active urinary tract infection.

PRIOR/CONCURRENT THERAPY:

At least 1 course of prior standard intravesical therapy required.

At least 4 weeks since intravesical treatment, with resolution of any local or systemic toxicity.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance status: ECOG 0 or 1.

Hematopoietic:

WBC at least 3,300;

Hemoglobin at least 10 g/dL.

Hepatic:

Bilirubin no greater than 1.5 mg/dL;

AST and ALT no greater than 2 times normal.

Renal: Creatinine no greater than 1.5 mg/dL.

OTHER:

Medically able to undergo cystoscopy.

No pregnant women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18
Dates: Start 1994-03; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Gansler T, Vaghmar N, Olson JJ, Graham SD. Suramin inhibits growth factor binding and proliferation by urothelial carcinoma cell cultures. J Urol. 1992 Sep;148(3):910-4. doi: 10.1016/s0022-5347(17)36776-9. PMID 1512858
- [Background] Walther MM, Figg WD, Linehan WM. Intravesical suramin: a novel agent for the treatment of superficial transitional-cell carcinoma of the bladder. World J Urol. 1996;14 Suppl 1:S8-11. doi: 10.1007/BF00182057. PMID 8738403
- [Background] Walther MM, Trahan EE, Cooper M, Venzon D, Linehan WM. Suramin inhibits proliferation and DNA synthesis in transitional carcinoma cell lines. J Urol. 1994 Nov;152(5 Pt 1):1599-602. doi: 10.1016/s0022-5347(17)32486-2. PMID 7933214